CLINICAL TRIAL: NCT07025967
Title: Using Mölkky for Community-dwelling Older Adults - A Pilot Randomized Controlled Trial
Brief Title: Using Mölkky for Community-dwelling Older Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, LIU Karen, Professor, The Hong Kong Polytechnic University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HongKongPU_Mölkky
Record Dates: First submitted 2025-06-10; First posted 2025-06-18 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-06

CONDITIONS: Older Adults Without Any Specific Clinical Condition
Keywords: Older adults; Physical activity; Physical functions; Cognitive functions; Well-being
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: A pilot study with a two-group, non-randomized controlled trial design
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mölkky group (Experimental): Participants will join the Mölkky.
  Interventions: Behavioral: Mölkky
- Home activity group (Active Comparator): Participants will receive home activities including closed-skilled exercises and cognitive training.
  Interventions: Behavioral: Home activity

INTERVENTIONS:
Behavioral: Mölkky — The Mölkky group participants receive two-hour weekly or bi-weekly Mölkky training sessions at their elderly community centers. In the sessions, participants are divided into two teams, taking turns throwing a wooden pin called the Mölkky to hit 12 smaller skittles. The fallen skittles are placed upright where they landed after each turn. The first team that reaches exactly 50 points wins.
  Arms: Mölkky group
Behavioral: Home activity — The participants in the home program receive weekly visits by social workers, physiotherapists, or occupational therapists at their homes for an activity regime including closed-skilled exercises and cognitive training. The closed-skilled exercises included stretching, elastic band exercises and functional exercises like tandem standing and bridging. Cognitive training included reality orientation, memory exercises, calculation, and mind-body exercises like Baduanjin.
  Arms: Home activity group

SUMMARY:
Physical activity is known to be a protector against major diseases. However, they usually do closed-skilled types, like jogging, swimming, Tai Chi. Our research showed that older adults benefit more from engaging in open-skilled activities. Mölkky is a Finnish throwing game that is considered an open-skilled activity.

The project investigates the benefits of Mölkky as an open-skilled physical activity and home activity for older adults.

DETAILED DESCRIPTION:
This study aims to examine the impacts of Mölkky on the overall functioning and psychological well-being of older adults when compared with a traditional home activity, including exercise and cognitive training.

45 older adults aged 60 or above from elderly service centres complete both baseline and post-program assessments. The Mölkky group receives Mölkky training in preparation for a Mölkky tournament, while the home activity group receives conventionally prescribed exercises and cognitive training. Assessments, including physical, cognitive, psychological and quality of life assessments, were conducted twice, at baseline and after 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* aged 60 or above,
* having no known pre-existing impairments that would prevent them from physical exercises, and
* had no known terminal disease leading to a life expectancy of less than one year.

Exclusion Criteria:

* cognitive impairment that makes them unable to complete the assessments, and
* a history of significant cardiovascular disease, respiratory disease or musculoskeletal dysfunction or exhibited steady hypertension (160/90 mmHg or above) that places them at risk of participating in an exercise program as determined by the centers

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Chinese Stroop Color and Word Test (Stroop) | Before the intervention to the end of intervention at 8 weeks; 6 months after the intervention
  The Chinese Stroop is used to assess participants' selective attention and cognitive flexibility. There are three sub-tests in the Stroop, identifying color of dots (Stroop I), identifying the words under incongruent conditions (Stroop II) and identifying the color of words under incongruent conditions (Stroop III). The time spent on each sub-test and errors which are not self-corrected are recorded. Time interference score is calculated by the formula: Interference = Stroop III - [(Stroop I + Stroop II) / 2], a lower time interference score indicates better performance. The Chinese Stroop has good reliability and validity.

SECONDARY OUTCOMES:
Hong Kong version of Montreal Cognitive Assessment (HK-MoCA) | Before the intervention to the end of intervention at 8 weeks; 6 months after the intervention
  The HK-MoCA is used to assess participants' overall cognitive ability including visuospatial function, naming, delayed recall, attention, language, abstraction, and orientation. A higher score out of 30 indicates better cognition. The HK-MoCA is a reliable and valid cognitive assessment.
Two-Minute Step Test (TMST) | Before the intervention to the end of intervention at 8 weeks; 6 months after the intervention
  The TMST is used to assess participants' lower limb muscle strength, endurance, and cardiorespiratory endurance. Participants are asked to repeat the action of stepping alternatively in two minutes, the total number of times the right knee is lifted is recorded. Post-it notes placed on the wall next to the participants are used as a height marker for each step, the greater the number of steps that meet the marker, the better the participants' cardiovascular fitness. The TMST is a reliable and valid assessment tool.
Timed Up and Go Test (TUG) | Before the intervention to the end of intervention at 8 weeks; 6 months after the intervention
  The TUG is used to assess participants' functional mobility. Participants are asked to stand up from a chair, walk 3 meters, turn around and go back to their seat. Time used is recorded, a shorter time indicates better physical functioning. The TUG is both reliable and valid assessment.
Geriatric Depression Scale Cantonese Version (GDS-C) | Before the intervention to the end of intervention at 8 weeks; 6 months after the intervention
  The GDS-C is used to assess participants' psychological well-being. Participants will answer 15 yes-no questions regarding their perception and attitude of their daily lives. A score of 8 or above indicates depressive symptoms. The GDS-C is reliable and valid.
EuroQol-five Dimensions Questionnaire - Hong Kong Chinese version (EQ-5D-5L) | Before the intervention to the end of intervention at 8 weeks; 6 months after the intervention
  The EQ-5D-5L is used to assess health-related QoL. Participants will rate their health states from 1 to 5 (1 indicates no problem and 5 indicates extreme problems/unable to perform) based on the severity of their problems in 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The 5-levels of health states are converted to a utility value using a local value. The EQ-5D-5L is reliable and valid.

OTHER OUTCOMES:
Physical Activity Enjoyment Scale (PAES) | Before the intervention to the end of intervention at 8 weeks
  The PAES is used to assess participants' attitudes towards physical activity. Participants will rate eight bipolar items by the scale of 1 to 7 on enjoyment, emotion, and engagement level. The negative items (Items 1, 4, 5 and 7) are reverse coded, meaning that score of 1 will be changed to 7, 2 changed to 6, 3 changed to 5 and vice versa. A score of 4 will remain unchanged for these negative items. The sum of scores of items is calculated. A higher PAES score indicates a greater level of enjoyment in physical activity. The PAES is reliable and valid.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Liu, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
The project is considering applying for external funding. The IPD can be shared after the funding application announcement and after data collection.